CLINICAL TRIAL: NCT04204473
Title: Phase I, Open-label, Single-arm Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Preliminary Efficacy of TY-9591 Tablets in Advanced NSCLC Patients With Epidermal Growth Factor Receptor( EGFR) Positive Mutation
Brief Title: A Study of TY-9591 in Advanced Non-small Cell Lung Cancer(NSCLC) Patients With EGFR Positive Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1601101
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-12

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TY-9591 (Experimental): Find maximum tolerated dose of TY-9591 given orally. Escalating doses of TY-9591 starting at 20mg daily.
  Interventions: Drug: TY-9591(10mg,40mg) qd. po

INTERVENTIONS:
Drug: TY-9591(10mg,40mg) qd. po — Increased dose cohorts from low dose to MTD(20mg Cohort1, 40mg Cohort2, 80mg Cohort3,120mg Cohort4, 160mg Cohort5, 200mg Cohort6)
  Other Names: TY-9591

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of TY-9591, with dose-escalation stage and dose-expansion stage.

DETAILED DESCRIPTION:
* To define the maximum tolerated dose(MTD) and the recommended phase 2 dose (RP2D)
* To investigate the pharmacokinetic profile of TY-9591 and its metabolites after single then multiple doses of TY-9591 administered orally once daily
* To evaluate the anti-cancer activity of TY-9591 in NSCLC patients with EGFR mutation(ORR、PFS、DoR、DCR、and CBR)

ELIGIBILITY:
Inclusion Criteria:

1. 18-75years old, male or female.
2. Histological or cytological confirmation diagnosis of NSCLC
3. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
4. Life expectancy of at least 3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
6. Documentation of disease progression while on previous continuous treatment with first-line EGFR TKI; patients must have confirmation of tumor EGFR activating mutations (exon 19 del, or exon 21 ) and T790M mutation status
7. Adequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

   a.Neutrophils (absolute value) ≥ 1.5×10^9/L; b.Hemoglobin ≥ 90 g/L; c.Platelet ≥ 80×10^9/L; d.Serum total bilirubin ≤ 1.5× ULN（for Patients with Gilbert Syndrome, total bilirubin ≤ 3×ULN and bilirubin ≤ 1.5×ULN should be permitted） f. Aspartate aminotransferase(AST)、alanine aminotransferase(ALT) ≤ 2.5×ULN; for patients with hepatic metastases, AST、ALT ≤ 5×ULN; g. International standardized ratio (INR) < 1.5, and activated partial prothrombin time (APTT) < 1.5×ULN;
8. Female subjects have a negative urine or serum pregnancy.
9. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.

Exclusion Criteria:

1. Treatment with any of the following:

   1. Treatment with an EGFR TKI within 14 days or about 5x half-life, whichever is the longer, of the first dose of study drug;
   2. Any cytotoxic chemotherapy, investigational agents or anticancer drugs for the treatment from a previous treatment regimen within 4 weeks of the first dose of study treatment;
   3. Major surgery within 4 weeks of the first dose of study treatment;
   4. Radiotherapy with a limited field of radiation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation that had to be completed within 4 weeks of the first dose of study treatment;
   5. Previously treated by other third-generation epidermal growth factor receptor tyrosine kinase inhibitor(EGFR-TKI) for T790M (for example Osimertinib).
   6. Patients currently receiving (or at least within 1 week prior to receiving the first dose )medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 isoenzyme (CYP)3A4.
2. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
3. Spinal cord compression or brain metastases unless asymptomatic.
4. Dysphagia, or active digestive system diseases or previous significant bowel resection or medical conditions potentially affect TY-9591 absorption.
5. Cardiac function and disease are consistent with the following:

   1. Corrected QT interval(QTc)> 470 milliseconds from 3 electrocardiograms (ECGs);
   2. Any clinically important abnormalities in rhythm;
   3. Any factors that increase the risk of QTc prolongation;
   4. Left ventricular ejection fraction (LVEF) <50%;
6. Active human immunodeficiency virus (HIV), syphilis, hepatitis c virus (HCV) or hepatitis b virus (HBV) infection, with the exception of asymptomatic chronic hepatitis b or hepatitis c carriers.

7 .Previous history of interstitial lung disease(ILD)、drug-induced ILD or radiation pneumonitis require steroid treatment, or any evidence of clinically active ILD diseases.

8. Previous allogeneic bone marrow transplant. 9. Hypersensitivity to TY-9591 or similar compounds or excipients. 10.Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | First 29 days of dosing
  Incidence of Dose Limiting Toxicity (DLT)
Maximum Tolerated Dose (MTD) | 1year
  To determine the Maximum Tolerated Dose (MTD) of TY-9591 in subjects with NSCLC
Recommended Phase 2 dose (RP2D) | through study completion, an average of 2.5 years
  Recommended Phase 2 dose (RP2D) of TY-9591 in subjects with NSCLC
Overall Response Rate (ORR) | At least 24 weeks
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Cmax | pharmacokinetics(PK) blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12, 24, 48, 72,96,120,144,168 and 192 hours post-dose.
  Cmax of TY-9591 following single dose
Tmax | pharmacokinetics(PK) blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12, 24, 48, 72,96,120,144,168 and 192 hours post-dose.
  Tmax of TY-9591 following single dose
Area Under Curve(AUC) | pharmacokinetics(PK) blood samples are collected at pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10,12, 24, 48, 72,96,120,144,168 and 192 hours post-dose
  AUC of TY-9591 following single dose
Cmax | The datas should be evaluated multiple times on Cycle 1 day1,8,15, 21 pre-dose; Cycle 2 day1 (at pre-dose, 0.5,1, 2, 3, 4, 6, 8, 10,12, 24 hours post-dose). Each cycle is 21 days
  Cmax of TY-9591 following multiple dose
Cmin | The datas should be evaluated multiple times on Cycle 1 day1,8,15, 21 pre-dose; Cycle 2 day1 (at pre-dose, 0.5,1, 2, 3, 4, 6, 8, 10,12, 24 hours post-dose). Each cycle is 21 days
  Cmin of TY-9591 following multiple dose
AUC | The datas should be evaluated multiple times on Cycle 1 day1,8,15, 21 pre-dose; Cycle 2 day1 (at pre-dose, 0.5,1, 2, 3, 4, 6, 8, 10,12, 24 hours post-dose). Each cycle is 21 days
  AUC of TY-9591 following multiple dose
Progression-free survival (PFS) | 10.1 months
  PFS is defined as time from date of first dose of study treatment to date of first documented disease progression or death due to any cause determined by by Investigator assessment in accordance to RECIST 1.1
Duration of Response (DOR) | 9.7 months
  DOR is defined as the time from first documented response (PR or CR) to the date of first documented disease progression or death due to any cause determined by Investigator assessment in accordance to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No